CLINICAL TRIAL: NCT01029054
Title: Multicenter, Open-label, Single-arm, Phase 1b/2 Study of the Safety and Efficacy of Combination Treatment w/ Carfilzomib, Lenalidomide (Revlimid®) and Dexamethasone (CRD) in Subjects w/ Newly Diagnosed, Previously Untreated Multiple Myeloma Requiring Systemic Chemotherapy
Brief Title: Carfilzomib and Lenalidomide With Dexamethasone Combination in Newly Diagnosed, Previously Untreated Multiple Myeloma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: Onyx Therapeutics, Inc. (Industry); Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: UMCC 2009.056; HUM30396 (Other: University of Michigan Medical IRB)
Record Dates: First submitted 2009-12-08; First posted 2009-12-09 (Estimated); Results first posted 2014-11-20 (Estimated); Last update posted 2017-01-30 (Estimated); Status verified 2016-12

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — carfilzomib; Lenalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- carfilzomib, lenalidomide w/dexamethasone (Experimental): Phase I: carfilzomib will be taken with a combination of lenalidomide plus dexamethasone in a series of escalating dosages to determine the maximum tolerated dose level
  Phase II: carfilzomib will be given at the MTD established in the Phase I portion of the study
  Interventions: Drug: carfilzomib, lenalidomide plus dexamethasone

INTERVENTIONS:
Drug: carfilzomib, lenalidomide plus dexamethasone — Phase I: Carfilzomib will be administered at the dosage assigned for the subject's cohort as an IV infusion on Days 1, 2, 8, 9, 15, and 16 of a 28-day cycle for Cycles 1 - 8 (induction) and on Days 1, 2, 15, and 16 of a 28-day cycle for Cycles 9+ (maintenance).
  Lenalidomide will be administered PO daily at 25 mg on Days 1- 21 of the 28-day cycle for Cycles 1 - 8+.
  Dexamethasone 40 mg will be administered PO or IV between 30 minutes and 4 hours preceding the carfilzomib push.
Drug: carfilzomib, lenalidomide plus dexamethasone — Phase II: Carfilzomib will be administered at the Maximum Tolerated Dose (MTD) established in Phase I as an IV infusion on Days 1, 2, 8, 9, 15, and 16 of a 28-day cycle for Cycles 1 - 8 (induction) and on Days 1, 2, 15, and 16 of a 28-day cycle for Cycles 9+ (maintenance).
  Lenalidomide will be administered PO daily at 25 mg on Days 1- 21 of the 28-day cycle for Cycles 1 - 8+.
  Dexamethasone will be administered PO or IV between 30 minutes and 4 hours preceding the carfilzomib push on Days 1, 8, 15, and 22 as follows: Cycles 1-4: 40 mg; Cycles 5-8: 20 mg; and Cycles 9 and higher: 10 mg.

SUMMARY:
This study is designed to evaluate the safety and to determine the maximum tolerated dose of carfilzomib + lenalidomide in combination with dexamethasone in newly diagnosed Multiple Myeloma patients who have not received treatment.

DETAILED DESCRIPTION:
During the Phase I portion of this clinical trial, the dose of Revlimid® and carfilzomib will be increased until the best and safest amount (or dose) is identified in combination with standard doses of Revlimid® and dexamethasone. "Investigational" means that the drug combination is still being studied and that research doctors are trying to find out more about it such as the safest dose to use, the side effects it may cause and how effective the Revlimid® and carfilzomib and dexamethasone investigational combination is for treating newly diagnosed multiple myeloma. In this clinical trial we are looking for the highest dose of the combination that can be given safely and see how well it works as a combination in newly diagnosed patients.

The drug, carfilzomib, has not yet been approved by the FDA (U.S. Food and Drug Administration). Revlimid® and Dexamethasone have been approved by the FDA. The drugs have not been approved in this combination for use for your type of cancer or any other type of cancer. Carfilzomib is being researched to treat multiple myeloma. Dexamethasone is commonly used, either alone, or in combination with other drugs, to treat multiple myeloma. Revlimid® is currently approved by the US FDA in combination with dexamethasone for the treatment of patients with multiple myeloma who have received at least 1 prior therapy.

After the Phase I clinical trial defines the safest doses of Revlimid® and carfilzomib and dexamethasone that can be taken together, the research study will move on to its second portion, a Phase II clinical trial. The Phase II portion of the clinical trial will test the clinical effectiveness of the best dose combination of the three drugs.

ELIGIBILITY:
Inclusion Criteria

1. Newly diagnosed, histologically confirmed, previously untreated Stage I, II, or III multiple myeloma requiring systemic chemotherapy
2. Diagnosis of symptomatic multiple myeloma per IMWG uniform criteria within the past 90 days
3. Measurable disease, per IMWG (International Myeloma Working Group) criteria (>= one of the following) within the past 4 weeks:

   * Monoclonal protein >= 0.5 g/dL by serum protein electrophoresis
   * Monoclonal light chain >= 200 mg by 24-hour urine protein electrophoresis
   * If serum protein electrophoresis is felt to be unreliable for routine M-protein measurement, then quantitative immunoglobulin levels are acceptable
4. Life expectancy > 3 months
5. Eastern Cooperative Oncology Group (ECOG) performance status 0-2
6. Adequate hepatic function, with bilirubin < 1.5 x the ULN, and AST (Aspartate Aminotransferase) and ALT (Alanine Transaminase) < 2.5 x ULN
7. Absolute neutrophil count (ANC) >=1.0 x 109/L, hemoglobin >= 8 g/dL, platelet count >= 75 x 109/L
8. Calculated creatinine clearance (by Cockroft-Gault) >= 60 ml/min
9. Written informed consent in accordance with federal, local, and institutional guidelines.
10. Subjects must agree to adhere to all study requirements, including birth control measures and pregnancy testing, visit schedule, outpatient treatment, required concomitant medications, and laboratory monitoring.
11. Must be able to take either 81 mg or 325 mg aspirin daily as prophylactic anticoagulation.

Exclusion Criteria

1. Non-secretory or hyposecretory multiple myeloma, defined as <0.5 g/dL M-protein in serum, <200 mg/24 hr urine M-protein, or disease only measured by serum free light chain
2. POEMS (Polyneuropathy, Organomegaly, Endocrinopathy, Monoclonal Gammopathy, and Skin Changes) syndrome
3. Plasma cell leukemia
4. Waldenström's macroglobulinemia or IgM myeloma
5. Radiotherapy to multiple sites or immunotherapy within 2 weeks before start of protocol treatment (localized radiotherapy to a single site at least 1 week before start is permissible)
6. Patient must not have been previously treated with any prior systemic therapy for the treatment of multiple myeloma

   * Prior treatment of hypercalcemia or spinal cord compression or aggressively progressing myeloma with corticosteroids does not disqualify the patient (the dose should not exceed the equivalent of 160 mg of dexamethasone in a 2 week period)
   * Bisphosphonates are permitted
7. Participation in an investigational therapeutic study within 3 weeks or within 5 drug halflives (t1/2) prior to first dose, whichever time is greater
8. Pregnant or lactating females
9. History of allergy to mannitol
10. Major surgery within 3 weeks prior to first dose
11. Myocardial infarction within 3 months prior to enrollment, NYHA (New York Heart Association) Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities
12. Uncontrolled hypertension or diabetes
13. Acute active infection requiring systemic antibiotics, antivirals, or antifungals within two weeks prior to first dose
14. Known or suspected HIV infection, known HIV seropositivity
15. Active hepatitis infection
16. Non-hematologic malignancy within the past 3 years except a) adequately treated basal cell, squamous cell skin cancer, thyroid cancer, carcinoma in situ of the cervix, or prostate cancer < Gleason Grade 6 with stable prostate specific antigen levels or cancer considered cured by surgical resection alone
17. Any clinically significant medical disease or condition that, in the Investigator's opinion, may interfere with protocol adherence or a subject's ability to give informed consent
18. Significant neuropathy (Grade >2) at the time of the first dose and/or within 14 days before enrollment
19. Contraindication to any of the required concomitant drugs
20. Subjects in whom the required program of PO and IV fluid hydration is contraindicated
21. Subjects with known or suspected amyloidosis of any organ
22. Subjects with pleural effusions requiring thoracentesis or ascites requiring paracentesis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2009-09; Primary Completion 2011-12 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Kaminski, M.D., Principal Investigator — University of Michigan Rogel Cancer Center
Locations (4):
- United States (4):
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Mt. Sinai Medical Center, New York, New York

REFERENCES:
- [Derived] Landgren O, Kazandjian D, Roussel M, Jasielec J, Dytfeld D, Anderson A, Kervin TA, Iskander K, McFadden I, Jakubowiak AJ. Efficacy and safety of carfilzomib-lenalidomide-dexamethasone in newly diagnosed multiple myeloma: pooled analysis of four single-arm studies. Leuk Lymphoma. 2022 Oct;63(10):2413-2421. doi: 10.1080/10428194.2022.2068001. Epub 2022 May 12. PMID 35549810
- [Derived] Jakubowiak AJ, Dytfeld D, Griffith KA, Lebovic D, Vesole DH, Jagannath S, Al-Zoubi A, Anderson T, Nordgren B, Detweiler-Short K, Stockerl-Goldstein K, Ahmed A, Jobkar T, Durecki DE, McDonnell K, Mietzel M, Couriel D, Kaminski M, Vij R. A phase 1/2 study of carfilzomib in combination with lenalidomide and low-dose dexamethasone as a frontline treatment for multiple myeloma. Blood. 2012 Aug 30;120(9):1801-9. doi: 10.1182/blood-2012-04-422683. Epub 2012 Jun 4. PMID 22665938

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Escalation Cohort 1: Carfilzomib will be administered as an IV infusion on Days 1, 2, 8, 9, 15, and 16 of a 28-day cycle for Cycles 1 - 8 (induction) and on Days 1, 2, 15, and 16 of a 28-day cycle for Cycles 9+ (maintenance) at dose level 20 mg/m^2.
  Lenalidomide will be administered PO daily at 25 mg on Days 1- 21 of the 28-day cycle for Cycles 1 - 8+.
  Dexamethasone will be administered PO or IV between 30 minutes and 4 hours preceding the carfilzomib push.
- Dose Escalation Cohort 2: Carfilzomib will be administered as an IV infusion on Days 1, 2, 8, 9, 15, and 16 of a 28-day cycle for Cycles 1 - 8 (induction) and on Days 1, 2, 15, and 16 of a 28-day cycle for Cycles 9+ (maintenance) at dose level 27 mg/m^2.
  Lenalidomide will be administered PO daily at 25 mg on Days 1- 21 of the 28-day cycle for Cycles 1 - 8+.
  Dexamethasone will be administered PO or IV between 30 minutes and 4 hours preceding the carfilzomib push.
- Dose Escalation Cohort 3: Carfilzomib will be administered as an IV infusion on Days 1, 2, 8, 9, 15, and 16 of a 28-day cycle for Cycles 1 - 8 (induction) and on Days 1, 2, 15, and 16 of a 28-day cycle for Cycles 9+ (maintenance) at dose level 36 mg/m^2.
  Lenalidomide will be administered PO daily at 25 mg on Days 1- 21 of the 28-day cycle for Cycles 1 - 8+.
  Dexamethasone will be administered PO or IV between 30 minutes and 4 hours preceding the carfilzomib push.
Period: Phase I
Arm/Group | Dose Escalation Cohort 1 | Dose Escalation Cohort 2 | Dose Escalation Cohort 3
Started | 4 | 13 | 18
Completed | 4 | 13 | 18
Not Completed | 0 | 0 | 0
Period: Phase II
Arm/Group | Dose Escalation Cohort 1 | Dose Escalation Cohort 2 | Dose Escalation Cohort 3
Started | 0 | 0 | 18 (35 participants were enrolled in Ph I. 18 additional participants were enrolled in Ph II at the MTD.)
Completed | 0 | 0 | 18
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Carfilzomib, Lenalidomide w/Dexamethasone: Carfilzomib will be administered as an IV infusion on Days 1, 2, 8, 9, 15, and 16 of a 28-day cycle for Cycles 1 - 8 (induction) and on Days 1, 2, 15, and 16 of a 28-day cycle for Cycles 9+ (maintenance).
  Lenalidomide will be administered PO daily at 25 mg on Days 1- 21 of the 28-day cycle for Cycles 1 - 8+.
  Dexamethasone will be administered PO or IV between 30 minutes and 4 hours preceding the carfilzomib push.
Arm/Group | Carfilzomib, Lenalidomide w/Dexamethasone
Number analyzed (Participants) | 53
Age, Continuous [Median (Full Range); unit: years] | 59 [35 to 81]
Gender [Count of Participants; unit: Participants]
  Female | 14
  Male | 39

OUTCOME MEASURES:

1. Primary Outcome: The Maximum Tolerated Dose (MTD) of Carfilzomib
Description: Determine the MTD of Carfilzomib when combined with Lenalidomide and Dexamethasone. The estimated time to determine the MTD is 6 months.
Time Frame: 6 Months
Population: Of the 53 patients enrolled, 35 were entered into the Phase I portion of the study.
Measure: Number; unit: mg/m^2
Arm/Group | Carfilzomib, Lenalidomide w/Dexamethasone
Number analyzed (Participants) | 35
mg/m^2 | 36

2. Secondary Outcome: The Percentage of Patients Alive Without Progression
Description: The Progression Free Survival (PFS) rate will be determined at 12 and 24 months post treatment.
  Progressive Disease (PD) is defined as an increase of greater than or equal to 25% from lowest response level in serum M-component and/ or urine M-component and/ or the difference between involved or uninvolved SFLC levels and/ or bone marrow % plasma cells. PD may also be the development of new bone lesions or soft tissue plasmacytomas or the increase in size of existing lesions. PD may also be the development of hypercalcemia.
Time Frame: 12 Months and 24 Months Post Treatment
Measure: Number; unit: percentage of patients
Arm/Group | Carfilzomib, Lenalidomide w/Dexamethasone
Number analyzed (Participants) | 53
percentage of patients
  Percentage of Patients Without Progression at 12 m | 97
  Percentage of Patients Without Progression at 24 m | 92

3. Primary Outcome: The Percentage of Patients That Achieve a Response to Treatment
Description: The percentage of patients that achieve at least a sCR (Stringent Complete Response), at least a VGPR (Very Good Partial Response) and at least a PR (Partial Response) will be determined.
  sCR is defined as:
  * Negative immunofixation on the serum and urine and
  * Disappearance of any soft tissue plasmacytomas and
  * < 5% plasma cells in bone marrow and
  * Normal SFLC ratio and
  * Absence of clonal cells in bone marrow
  VGPR is defined as:
  * Serum and urine M-protein detectable by immunofixation but not on electrophoresis or
  * ≥ 90% reduction in serum M-component with urine M-component < 100 mg per 24 hours
  PR is defined as:
  * ≥ 50% reduction of serum M-protein and reduction in 24-hour urinary M-protein by ≥ 90% or to < 200 mg per 24 hours
  * If present at baseline, a ≥ 50% reduction in the size of soft tissue plasmacytomas is also required
Time Frame: 4 Months After Treatment Start
Measure: Number; unit: percentage of patients
Arm/Group | Carfilzomib, Lenalidomide w/Dexamethasone
Number analyzed (Participants) | 53
percentage of patients
  % of patients that achieve at least a sCR | 42
  % of patients that achieve at least a VGPR | 81
  % of patients that achieve at least a PR | 98

ADVERSE EVENTS:
Time Frame: All Adverse Events (AEs) that occurred after the subject signed consent were documented.
Description: A Serious Adverse Event (SAE) is defined as: death, a life-threatening experience, hospitalization, results in persistent or significant disability/incapacity, congenital anomaly/birth defect in the offspring of an exposed subject, important medical events based upon appropriate medical judgment, pregnancy.
Arm/Group | Carfilzomib, Lenalidomide w/Dexamethasone
Serious Adverse Events (participants affected / at risk) | 23/53
Other Adverse Events (participants affected / at risk) | 53/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Carfilzomib, Lenalidomide w/Dexamethasone (N=53)
Acute Renal Failure (Renal and urinary disorders) | 2
Acute Mental Status Change (Nervous system disorders) | 1
Appendicitis (Infections and infestations) | 1
Atrial Fibrillation (Cardiac disorders) | 1
Clostridium Difficile (Infections and infestations) | 1
Colitis (Gastrointestinal disorders) | 1
Compression Fracture (Musculoskeletal and connective tissue disorders) | 1
Confusion (Nervous system disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Febrile Neutropenia (Blood and lymphatic system disorders) | 1
Fever (General disorders) | 1
Gastroenteritis (Gastrointestinal disorders) | 1
Grand Mal Seizure (Nervous system disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 2
Pneumonia (Infections and infestations) | 4
Influenza (Infections and infestations) | 1
Anemia (Blood and lymphatic system disorders) | 2
Intracranial Hemorrhage (Vascular disorders) | 1
Methemoglobinemia (Blood and lymphatic system disorders) | 1
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary Toxicity (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1
Rapid Ventricular Response (Cardiac disorders) | 1
Seizure (Nervous system disorders) | 1
Urinary Tract Infection (Infections and infestations) | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Carfilzomib, Lenalidomide w/Dexamethasone (N=53)
Hyperglycemia (Metabolism and nutrition disorders) | 38
Edema (General disorders) | 25
Hypophosphatemia (Metabolism and nutrition disorders) | 24
Fatigue (General disorders) | 20
Muscle Cramping (Musculoskeletal and connective tissue disorders) | 17
Rash (Skin and subcutaneous tissue disorders) | 15
Elevated Liver Function Test (Investigations) | 15
Diarrhea (Gastrointestinal disorders) | 14
Infection (Infections and infestations) | 12
Phlebitis (Vascular disorders) | 12
Peripheral Neuropathy (Nervous system disorders) | 12
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8
Deep Vein Thrombosis (Vascular disorders) | 6
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 3
Nausea (Gastrointestinal disorders) | 7
Renal (Renal and urinary disorders) | 5
Constipation (Gastrointestinal disorders) | 5
Mood Alterations (Psychiatric disorders) | 5
Thrombocytopenia (Blood and lymphatic system disorders) | 36
Anemia (Blood and lymphatic system disorders) | 32
Neutropenia (Blood and lymphatic system disorders) | 16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes